CLINICAL TRIAL: NCT01261273
Title: Prospective, Single-Arm, Multi-Centre, Observational Registry to Further Validate Safety and Efficacy of the Nobori DES in Real-World Patients
Brief Title: e-NOBORI Observational Registry of Nobori DES
Acronym: e-NOBORI
Status: Completed | Type: Observational
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Other Study IDs: T113E2
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Coronary Artery Disease
Keywords: PCI; observational registry
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (14):
- Stable angina: Patient admitted with stable angina
- Acute Coronary Syndrome: Patients admitted with Acute Coronary Syndrome
- Female: Participant female patients
- Bifurcation: One or more lesions treated during the baseline in bifurcation
- Insulin Dependent Diabetes Mellitus: Patients that were insulin-dependent diabetes mellitus at admission
- Non-Insulin Dependent Diabetes Mellitus: Patients that were non-insulin-dependent diabetes mellitus at admission
- Small Vessels: vessels smaller or equal to 2.75mm
- NOBORI Long Lesions: Lesions longer or equal to 20mm
- Renal Insufficiency: Patients that at admission had renal insufficiency (> 2.0 mg/dL - 176 µmol/mL) at admission
- Elderly: Patients more or equal 80 years old
- Restenosis: One or more lesions treated during the baseline in were restenotic lesions
- Multivessel Treatment: Patients who underwent the treatment of more than 1 vessel during the index procedure
- Complex Lesions: Patients who underwent a PCI on the Left Main Trunk, on a Chronic Total Occluded lesion or located on a Saphenous Vein Graft
- Overall: Total Population

SUMMARY:
Title Prospective, single-arm, multi-centre, observational registry to further validate safety and efficacy of the Nobori® DES in real-world patients.

Objective Primary objective The primary objective of e-NOBORI registry is to further validate the safety and efficacy of Nobori® DES system in unselected patients representing everyday clinical practice.

Primary Endpoint: Freedom from Target Lesion Failure (TLF) defined as a composite of cardiac death, target vessel related myocardial infarction (MI) and clinically driven target lesion revascularization (TLR) at 1 year

DETAILED DESCRIPTION:
* Title Prospective, single-arm, multi-centre, observational registry to further validate safety and efficacy of the Nobori® DES in real-world patients.
* Primary objective The primary objective of e-NOBORI registry is to further validate the safety and efficacy of Nobori® DES system in unselected patients representing everyday clinical practice.
* Primary Endpoint: Freedom from Target Lesion Failure (TLF) defined as a composite of cardiac death, target vessel related myocardial infarction (MI) and clinically driven target lesion revascularization (TLR) at 1 year
* Clinical Site Locations:

Up to 200 centres across Europe, Asia and Central and South America

-Patient Population : ~18000 eligible patients suitable for treatment with the Nobori® DES will be entered in the e-NOBORI registry

Eligibility Criteria

* Patient is more or equal 18 years old;
* Patient is, according to hospital routine practice, eligible for percutaneous coronary intervention using DES (and RVD matches available Nobori® DES sizes);
* Patient has been informed of the nature of the study and agrees to its provisions, has provided written informed consent as approved by the Institutional Review Board/Ethics Committee of the respective clinical site, wherever such requirement exists.

NOTE: In order to avoid bias it is recommended that all investigators aim to enrol all consecutive patients complying with study eligibility criteria. It is also desirable to have at least two cardiologists as investigators in each centre.

According to pre-specified criteria, patients will be automatically allocated to one or more sub-studies as following:

* NOBORI Acute Coronary Syndrome
* NOBORI Stable angina
* NOBORI Female
* NOBORI Bifurcation
* NOBORI Diabetes

  * Insulin Dependent Diabetes Mellitus (IDDM)
  * Non-Insulin Dependent Diabetes Mellitus (NIDDM)
* NOBORI Small Vessels (less or equal 2.75mm)
* NOBORI Long Lesions (more or equal 20mm)
* NOBORI Renal Insufficiency (> 2.0 mg/dL - 176 µmol/mL)
* NOBORI Elderly (more or equal 80 years of age)
* NOBORI Restenosis
* NOBORI Multivessel Treatment
* NOBORI Complex Lesions

In addition to above mentioned sub-studies there will be geographic sub-studies for the main areas.

Medication Pre-Procedure: According to hospital routine practice Post-Procedure: Mandatory antiplatelet treatment, according to hospital routine practice (minimum 6 months DAT)

ELIGIBILITY:
Inclusion Criteria:

* Patient is more or equal 18 years old;
* Patient is, according to hospital routine practice, eligible for percutaneous coronary intervention using DES (and RVD matches available Nobori® DES sizes);
* Patient has been informed of the nature of the study and agrees to its provisions, has provided written informed consent as approved by the Institutional Review Board/Ethics Committee of the respective clinical site, wherever such requirement exists.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suitable for PCI intervention
Sampling Method: Probability Sample
Enrollment: 18000 (Actual)
Dates: Start 2010-08-25 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05-27 (Actual)

PRIMARY OUTCOMES:
FREEDOM OF TARGET LESION FAILURE | 1 YEAR
  TLF: COMPOSITE OF CARDIAC DEATH, MYOCARDIAL INFARCTION AND TARGET LESION REVASCULARIZATION

SECONDARY OUTCOMES:
Procedural success | 1 MONTH
  Procedural success is defined as achievement of a diameter of stenosis of <30% by visual assessment and/or <50% by QCA, using any percutaneous method, without the occurrence of death, MI, or repeat revascularization of the target lesión during the hospital stay.
Device success | 1 MONTH
  Device Success defined as attainment of a final residual diameter stenosis of the target lesion of < 30% by visual assessment and/or < 50% by QCA, using the assigned device only.
  Device Success defined as attainment of a final residual diameter stenosis of the target lesion of < 30% by visual assessment and/or < 50% by QCA, using the assigned device only.
  Device success is defined as attainment of a final residual diameter stenosis of the target lesión of <30% by visual assessment and/or >50% QCA, using the assigned device only.
Acute/subacute stent thrombosis | 1 MONTH
  (definite/probable according to ARC definitions)
Peri-procedural myocardial infarction | 1 MONTH
  Peri-procedural myocardial infarction
Rate of Major Adverse Cardiac Events (MACE) | 1 MONTH
  Major Adverse Cardiac Events (MACE) defined as a composite of cardiac death, MI or clinically driven target vessel revascularization (TVR)
Major vascular and bleeding complications | 1 MONTH
  NOT CABG RELATED
Cardiac death/ Myocardial Infarction | 1 AND 2 YEARS
  Cardiac death/ Myocardial Infarction
Clinically driven target lesion revascularization (TLR) | 1 & 2 YEARS
  re-PCI or CABG involving target lesion
Stent thrombosis | 1 AND 2 YEARS
  (definite/probable; ARC definition)
Clinically driven target vessel revascularization (TVR) | 1 AND 2 YEARS
  PCI AND CABG
Target Lesion Failure (TLF) | 1 MONTH AND 2 YEARS
  Defined as a composite of cardiac death, target vessel related myocardial infarction (MI) and clinically driven target lesion revascularization
Patient Oriented Composite Endpoint defined as any cause of mortality, MI (Q-wave and non Q-wave), or any TVR | 1 MONTH, 1 AND 2 YEARS
  Patient Oriented Composite Endpoint defined as any cause of mortality, MI (Q-wave and non Q-wave), or any TVR
Composite Endpoint of Cardiac death and MI | 1 MONTH, 1 AND 2 YEARS
  Composite Endpoint of Cardiac death and MI
Composite Endpoint of Cardiac death and post-procedural MI | 1 month, 1 and 2 years post-procedure
  Composite Endpoint of Cardiac death and post-procedural MI
Stent thrombosis | 1 month, 1 and 2 years post-procedure
  definite and probable according to ARC definitions
Primary Stent thrombosis | 1 month, 1 and 2 years post-procedure
  definite and probable according to ARC definitions
Secondary Stent thrombosis | 1 month, 1 and 2 years post-procedure
  definite and probable according to ARC definitions
Duration of dual antiplatelet therapy | UP TO 2 YEARS
  Duration of dual antiplatelet therapy
Composite Endpoint of Cardiac death, post-procedural MI and stent thrombosis rate during the course of DAT versus the same events after cessation of DAT | UP TO 2 YEARS
  Composite Endpoint of Cardiac death, post-procedural MI and stent thrombosis rate during the course of DAT versus the same events after cessation of DAT
Clinically driven Target Lesion Revascularization | 1 MONTH
  Clinically driven Target Lesion Revascularization
Clinically driven Target Vessel Revascularization | 1 MONTH
  Clinically driven Target Vessel Revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Dragica Paunovic, Dr., Study Chair — Terumo Europe
Locations (257):
- SMZ-Donauspital Vienna, Vienna, Austria
- National Heart Foundation Hospital & Research Institute, Dhaka, Bangladesh
- Belarus (3):
  - Republican Clinical Medical Center (Presidential Hospital), Minsk
  - Republican Scientific and Practical Center of Cardiology, Minsk
  - Mogilev Regional Clinical Hospital, Mogilev
- Brazil (32):
  - Hospital Madre Teresa, Belo Horizonte
  - Hospital Santa Isabel-Sociedade Divina Providência, Blumenau
  - HMCP PUC-Campinas, Campinas
  - Hospital E Maternidade Madre Teodora, Campinas
  - Hospital Vera Cruz Campinas, Campinas
  - Hospital Geral Universitário, Cuiabá
  - Hospital Cruz Vermelha Brasileira Filial do Paraná, Curitiba
  - Hospital Nossa Senhora das Graças, Curitiba
  - Hospital Santa Cruz, Curitiba
  - Hospital Monte Sinai (Juiz de Fora), Juiz de Fora
  - Instituto Cardiovascular de Linhares (Unicor), Linhares
  - Hospital do Coração de Londrina, Londrina
  - Hospital Paraná, Maringá
  - Irmandade da Santa Casa de Misericórdia de Marília, Marília
  - Hospital Procordis, Niterói
  - Hospital Vera Cruz Patos de Minas, Patos de Minas
  - Hospital Moinhos de Vento, Porto Alegre
  - Hospital Mãe De Deus, Porto Alegre
  - Hospital São Lucas - PUCRS, Porto Alegre
  - Clinica Status Cor, Rio de Janeiro
  - Hospital Naval Marcíllo Dias, Rio de Janeiro
  - Fundação Bahiana de Cardiologia (MC Oliveira Prest, Salvador
  - Hospital Beneficencia Portuguesa de Sao Paulo, São João do Paraíso
  - Casa de Saude Santa Marcelina, São Paulo
  - Hospital Albert Einstein, São Paulo
  - Hospital Bandeirantes, São Paulo
  - Instituto Dante Pazzanese, São Paulo
  - Real e Benemérita Assoção Portuguesa de Beneficênc, São Paulo
  - Hospital Ana Costa (ENDOCOR Serviços Médicos Ltda), São Vicente
  - Hospital Anchieta Ltda., Taguatinga
  - Instituto do Coração do Triângulo Mineiro, Uberlândia
  - Insituto de Cardiologia Espirito Santo, Vitória
- Tokuda Hospital Sofia, Sofia, Bulgaria
- Chile (7):
  - Hospital Militar de Santiago, La Reina
  - clinica Santa Maria, Santiago
  - Instituto Nacional del Torax, Santiago
  - San Juan de Dios, Santiago
  - Las Higueras De Talcahuano, Talcahuano
  - V Region (Hospital Gustavo Fricke, Hospital Van Buren, Clinica Reñaca), Valparaíso
  - Clinica alemana de Santiago, Vitacura
- Czechia (2):
  - St. Anne University Hospital, Brno
  - Nemocnice Na Homolce, Prague
- Gentofte Hospital (M12FU), Hellerup, Denmark
- Egypt (16):
  - Glory cardiac center - Cath group, Al Mansurah
  - ALHYATT Cardiovascular Center, Alexandria
  - International Cardiac Center, Alexandria
  - AL Amal, Cairo
  - Al Nakhil hospital, Cairo
  - AS-Salam Mohndseen, Cairo
  - Cleopatra, Cairo
  - Egyheart - cath lab, Cairo
  - El Dorah Heart Care Center, Cairo
  - Hayat Hospital, Cairo
  - (DAFH) Dar Al Fouad Hospital, Giza
  - Alfa, Giza
  - ICS center, Giza
  - RCC Cardiac center, Giza
  - Al Noor Cath Lab, Sohag
  - Om El kora cardiac center, Tanta
- Estonia (2):
  - East Tallinn Central Hospital, Tallinn
  - North-Estonia Regional Hospital, Tallinn
- France (53):
  - Clinique de l'Europe à Amiens (SAS Cardio Amiens), Amiens
  - CHU Angers, Angers
  - Hôpital Privé d'Antony, Antony
  - Hopital La Roseraie, Aubervilliers
  - CH Avignon, Avignon
  - Clinique Rhone Durance, Avignon
  - CH Bastia, Bastia
  - Clinique La Fourcade, Bayonne
  - Clinique Bois Bernard à Bois Bernard, Bois-Bernard
  - Clinique Saint Augustin, Bordeaux
  - CHU de la Cavale Blanche, Brest
  - CH Privé Saint - Martin Caen, Caen
  - CHU de la Cote de Nacre (CHU Caen), Caen
  - Hopital Albert Schweitzer-Colmar, Colmar
  - CH Sud Francilien, Corbeil-Essonnes
  - Clinique des Cèdres-Dr Brunelle, Cornebarrieu
  - Clinique des Cèdres-Dr.Tauzin, Cornebarrieu
  - Centre Cardiologique d'Evecquemont, Évecquemont
  - CH Haguenau, Haguenau
  - CH de Lagny-Marne La Vallée, Jossigny
  - CH de Cornouaille, La Cornuaille
  - CH La Roche sur Yon, La Roche-sur-Yon
  - CH de Chartres, Le Coudray
  - CC Marie Lannelongue, Le Plessis-Robinson
  - Clinique La Louviere, Lille
  - CH Dupuytren Limoges, Limoges
  - CH Lorient, Lorient
  - Institut Hospitalier Jacques Cartier (ICPS Massy), Massy
  - Clinique les Fontaines, Melun
  - Clinique du Millenaire, Montpellier
  - Association Clinique Bizet, Paris
  - Clinique Turin - Paris, Paris
  - Hopital Lariboisière, Paris
  - Hopital Pitié Salpétrière, Paris
  - Hôpital du Val de Grâce, Paris
  - Hôpital Europeen Georges Pompidou (HEGP), Paris
  - CH Pau, Pau
  - CH Général Maréchal Joffre Perpignan, Perpignan
  - Clinique Saint-Martin Pessac, Pessac
  - CH Périgueux, Périgueux
  - CHU La Miletrie Poitiers, Poitiers
  - CH René Dubos, Pontoise
  - Hopital Claude Galien, Quincy
  - Clinique Saint Laurent, Rennes
  - Hôpital Jacques Puel (CH de Rodez), Rodez
  - Clinique Saint Hilaire, Rouen
  - Centre Cardiologique du Nord, Saint-Denis
  - NHC Strasbourg, Strasbourg
  - Clinique de l'Ormeau - CCV des Pyrenées, Tarbes
  - Polyclinique du Parc Toulouse, Toulouse
  - CH Valence, Valence
  - Clinique Vauban, Valenciennes
  - CH Bretagne Atlantique, Vannes
- JoAnn Medical Center, Tbilisi, Georgia
- Germany (18):
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Herz-und Diabeteszentrum Nordrhein-Westfalen, Bad Oeynhausen
  - Evangelisch Freikirchliches Krankenhaus und Herzze, Berlin
  - Gemeinschaftskrankenhaus Havelhöhe, Berlin
  - Jüdisches Krankenhaus, Berlin
  - Klinikum Neukölln, Berlin
  - Vivantes Klinkum Spandau, Berlin
  - Vivantes Netzwerk für Gesundheit gmbH - Am Urban, Berlin
  - Vivantes Netzwerk für Gesundheit gmbH - Friedrichs, Berlin
  - Vivantes Netzwerk für Gesundheit gmbH - Humboldt, Berlin
  - Ev.Bethesda-Johanniter Klinikum Duisburg GmbH, Duisburg
  - Klinikum Fulda, Fulda
  - Uniklinik Schleswig-Holstein, Campus Kiel, Kiel
  - Herzzentrum Leipzig-Rhöne Klinikum, Leipzig
  - St. Marienhospital Lünen, Lünen
  - Klinikum Oldenburg, Oldenburg
  - Universitätsklinik Rostock, Rostock
  - Evang.Diakonieanstalt Speyer, Speyer
- Hungary (3):
  - Gottsegen National Cardiology Institute (GOKI), Budapest
  - Semmelweis University Cardiology Centre, Budapest
  - Fejér Megyei Szent György Kórház, Székesfehérvár
- Indonesia (3):
  - Medistra Hospital, Jakarta
  - National Cardiovascular Center Harapan Kita, Jakarta
  - Dr. Soetomo General Hospital, Surabaya, Surabaya
- Ireland (2):
  - Beaumont Hospital, Dublin
  - University Hospital Galway, Galway
- Israel (6):
  - Rambam Medical centre, Haifa
  - Wolfson Medical Center, Holon
  - Meir Medical Center, Kfar-Saba, Kfar Saba
  - Laniado Medical Center, Netanya
  - Rabin Medical Center, Petah Tikva
  - Kaplan Hospital, Rehovot
- Latvia (2):
  - Invasive Cardiology Laboratory of Clinics "Gailezers" of Riga's Eastern Clinical University Hospital, Riga
  - Invasive Cardiology Laboratory of P. Stradins Clinical University Hospital, Riga
- Hospital of Lithuania University of Health Science, Kaunas, Lithuania
- Mater Dei, Msida, Malta
- Mexico (12):
  - Hospital Angeles Culiacan, Culiacán
  - Hospital Angeles Leon, León, Guanajuato
  - Hospital Star Medica Mérida Yucatán, Merida, Yucatan
  - 1e de Octubre ISSSTE, Mexico City
  - Centro Médico Nacional 20 de Noviembre, Mexico City
  - Hospital Angeles Mocel, Mexico City
  - Hospital Central Militar, Mexico City
  - Hospital de Cardiologia C.M.N., Mexico City
  - Instituto Nacional De Cardiologia "Ignacio Chávez", Mexico City
  - Dalinde Medical Center, México, DF
  - Hospital Universitario Dr. José Eleuterio Gonzalez, Monterrey, Nuevo León
  - Hospital Lomas de San Luis Internacional, San Luis Potosi SLP
- Netherlands (4):
  - Amphia Hospital, Breda
  - Albert Schweitzer Hospital, Dordrecht
  - Jeroen Bosch Ziekenhuis, s'Hertogenbosch
  - Medisch Centrum Haaglanden, The Hague
- Poland (3):
  - St Adalbert Speciality Hospital, Gdansk
  - Szpital Klinicznk Przemienienia (University Hospital), Poznan
  - Szpital Wojewodzski Poznaniu, Poznan
- Cardiolife Hospital Timisoara, Timișoara, Romania
- Russia (12):
  - Chelyabinsk Regional Clinical Hospital, Chelyabinsk
  - Military Hospital N3 named by Vishnevsky, Krasnogorsk
  - State cardiovascular center based on regional clin, Krasnoyarsk
  - Regional Clinical Hospital, Kursk
  - Central Clinical Hospital N°2 Russia Railways, Moscow
  - Academian E.N Meshalkin State Research Institute of circulation Pathology, Novosibirsk
  - Federal cardiosurgerical center, Penza, Penza
  - Kirochnaya str.41, Saint Petersburg
  - Federal center of heart,blood and endocrinology diseases named by Almazov, Saint Petersburg
  - Saratov Research Institute of science for cardiology, Saratov
  - Regional Vessel Center, Ufa
  - Ufa city Emergency Hospital, Ufa
- Serbia (3):
  - Institute for Cardiovascular Disease Dedinje, Dedinje
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center of Niš, Niš
- CH Celje, Celje, Slovenia
- Spain (32):
  - Hospital Juan Canalejo, A Coruña
  - Hospital San Rafael, A Coruña
  - Hospital general de Albacete, Albacete
  - Hospital San Juan, Alicante
  - Hospital Torrecárdenas, Almería
  - Hospital G. Trias i Pujol, Badalona
  - Hospital Bellvitge, Barcelona
  - Hospital Sant Pau, Barcelona
  - Hospital de Cruces-Barakaldo, Bilbao- Vizcaya
  - Hospital de Galdakao, Bizkaia
  - Hospital Nostra Señora Rossell, Cartagena
  - Hospital General de Castellón, Castellon
  - Hospital San Pedro de Alcantara-Caceres, Cáceres
  - Hospital Nostra Señora Alarcos, Ciudad Real
  - Hospital Cabueñes, Gijón
  - Hospital Universitario de Guadalajara, Guadalajara
  - Clinica San Roque, Las Palmas
  - Hospital de León, León
  - Clínica Moncloa, Madrid
  - Hospital Fundacion Alcorcon, Madrid
  - Hospital Puerta de Hierro, Majadahonda-Madrid
  - Hospital Virgen Arrixaca, Murcia
  - Universitario central de Asturias, Oviedo
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Candelaria, Santa Cruz de Tenerife
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Virgen Salud, Toledo
  - Clínico Universitario Valencia, Valencia
  - Hospital Manises, Valencia
  - Hospital Meixoeiro-MEDTEC, Vigo
  - Hospital Txagorritxu, Vitoria-Gasteiz
  - Hospital Miguel Servet, Zaragoza
- Sweden (4):
  - Falun Lasarett, Falun
  - University Hospital Linköping, Linköping
  - Uppsala Akademiska Sjukhus, Kardiologkliniken, Uppsala
  - Central Lasarettet i Västerås, Angio/PCI lab. Medi, Västerås
- Taiwan (7):
  - E-da Hospital/Kaohsiung, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung R.o.c.
  - Chi Mei Medical Center/Tainan, Tainan
  - National Cheng Kung University Hospital, Tainan
  - Cheng Hsin General Hospital / Taipei, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, VACRS, Taipei
- Ukraine (4):
  - Kharkov Regional Hospital, Kharkiv
  - Feofaniya, Kiev
  - Ukrainian Institute of Cardiology, Kiev
  - National Institute of Cardiovascular Surgery AMS, Kyiv
- United Kingdom (18):
  - Queen Elizabeth Birmingham, Birmingham
  - Royal Blackpool hospital (Lancashire Heart Centre), Blackpool
  - Royal Cornwall hospital, Cornwell
  - Castle Hill Hospital, Cottingham
  - Southern Health and Social Care Trust Craigavon Ar, Craigavon
  - Scunthorpe general hospital, District of North East Lincolnshire
  - Dorset county Hospital, Dorset
  - Eastbourne General, Eastbourne
  - Glenfield general hospital, Glenfield
  - Conquest Hospital Hastings, Hastings
  - Kettering General Hospital, Kettering
  - Northwick Park, London
  - Freeman Hospital, Newcastle upon Tyne
  - Royal Gwent Hospital, Newport
  - Fairfield General Hospital, North Manchester
  - Frimley Park Hospital NHS Foundation Trust, Surrey
  - Pinderfield General Hospital, Wakefield
  - New Cross Wolverhampton, Wednesfield

REFERENCES:
- [Background] Sigwart U, Puel J, Mirkovitch V, Joffre F, Kappenberger L. Intravascular stents to prevent occlusion and restenosis after transluminal angioplasty. N Engl J Med. 1987 Mar 19;316(12):701-6. doi: 10.1056/NEJM198703193161201. PMID 2950322
- [Background] Detre KM, Holmes DR Jr, Holubkov R, Cowley MJ, Bourassa MG, Faxon DP, Dorros GR, Bentivoglio LG, Kent KM, Myler RK. Incidence and consequences of periprocedural occlusion. The 1985-1986 National Heart, Lung, and Blood Institute Percutaneous Transluminal Coronary Angioplasty Registry. Circulation. 1990 Sep;82(3):739-50. doi: 10.1161/01.cir.82.3.739. PMID 2394000
- [Background] Holmes DR Jr, Holubkov R, Vlietstra RE, Kelsey SF, Reeder GS, Dorros G, Williams DO, Cowley MJ, Faxon DP, Kent KM, et al. Comparison of complications during percutaneous transluminal coronary angioplasty from 1977 to 1981 and from 1985 to 1986: the National Heart, Lung, and Blood Institute Percutaneous Transluminal Coronary Angioplasty Registry. J Am Coll Cardiol. 1988 Nov;12(5):1149-55. doi: 10.1016/0735-1097(88)92593-4. PMID 2971699
- [Background] Fischman DL, Leon MB, Baim DS, Schatz RA, Savage MP, Penn I, Detre K, Veltri L, Ricci D, Nobuyoshi M, et al. A randomized comparison of coronary-stent placement and balloon angioplasty in the treatment of coronary artery disease. Stent Restenosis Study Investigators. N Engl J Med. 1994 Aug 25;331(8):496-501. doi: 10.1056/NEJM199408253310802. PMID 8041414
- [Background] Serruys PW, de Jaegere P, Kiemeneij F, Macaya C, Rutsch W, Heyndrickx G, Emanuelsson H, Marco J, Legrand V, Materne P, et al. A comparison of balloon-expandable-stent implantation with balloon angioplasty in patients with coronary artery disease. Benestent Study Group. N Engl J Med. 1994 Aug 25;331(8):489-95. doi: 10.1056/NEJM199408253310801. PMID 8041413
- [Background] Morice MC, Serruys PW, Sousa JE, Fajadet J, Ban Hayashi E, Perin M, Colombo A, Schuler G, Barragan P, Guagliumi G, Molnar F, Falotico R; RAVEL Study Group. Randomized Study with the Sirolimus-Coated Bx Velocity Balloon-Expandable Stent in the Treatment of Patients with de Novo Native Coronary Artery Lesions. A randomized comparison of a sirolimus-eluting stent with a standard stent for coronary revascularization. N Engl J Med. 2002 Jun 6;346(23):1773-80. doi: 10.1056/NEJMoa012843. PMID 12050336
- [Background] Stettler C, Wandel S, Allemann S, Kastrati A, Morice MC, Schomig A, Pfisterer ME, Stone GW, Leon MB, de Lezo JS, Goy JJ, Park SJ, Sabate M, Suttorp MJ, Kelbaek H, Spaulding C, Menichelli M, Vermeersch P, Dirksen MT, Cervinka P, Petronio AS, Nordmann AJ, Diem P, Meier B, Zwahlen M, Reichenbach S, Trelle S, Windecker S, Juni P. Outcomes associated with drug-eluting and bare-metal stents: a collaborative network meta-analysis. Lancet. 2007 Sep 15;370(9591):937-48. doi: 10.1016/S0140-6736(07)61444-5. PMID 17869634
- [Background] Moses JW, Leon MB, Popma JJ, Fitzgerald PJ, Holmes DR, O'Shaughnessy C, Caputo RP, Kereiakes DJ, Williams DO, Teirstein PS, Jaeger JL, Kuntz RE; SIRIUS Investigators. Sirolimus-eluting stents versus standard stents in patients with stenosis in a native coronary artery. N Engl J Med. 2003 Oct 2;349(14):1315-23. doi: 10.1056/NEJMoa035071. PMID 14523139
- [Background] Holmes DR Jr, Leon MB, Moses JW, Popma JJ, Cutlip D, Fitzgerald PJ, Brown C, Fischell T, Wong SC, Midei M, Snead D, Kuntz RE. Analysis of 1-year clinical outcomes in the SIRIUS trial: a randomized trial of a sirolimus-eluting stent versus a standard stent in patients at high risk for coronary restenosis. Circulation. 2004 Feb 10;109(5):634-40. doi: 10.1161/01.CIR.0000112572.57794.22. PMID 14769686
- [Background] Grube E, Silber S, Hauptmann KE, Mueller R, Buellesfeld L, Gerckens U, Russell ME. TAXUS I: six- and twelve-month results from a randomized, double-blind trial on a slow-release paclitaxel-eluting stent for de novo coronary lesions. Circulation. 2003 Jan 7;107(1):38-42. doi: 10.1161/01.cir.0000047700.58683.a1. PMID 12515740
- [Background] Chevalier B, Serruys PW, Silber S, Garcia E, Suryapranata H, Hauptmann K, Wijns W, Schuler G, Fath-Ordoubadi F, Worthley S, Thuesen L, Meredith I, Bressers M, Nagai H, Paunovic D. Randomised comparison of Nobori, biolimus A9-eluting coronary stent with a Taxus(R), paclitaxel-eluting coronary stent in patients with stenosis in native coronary arteries: the Nobori 1 trial. EuroIntervention. 2007 Feb;2(4):426-34. PMID 19755281
- [Background] Ostojic M, Sagic D, Beleslin B, Jung R, Perisic Z, Jagic N, Nedeljkovic M, Mangovski L, Milosavljevic B, Stojkovic S, Orlic D, Antonic Z, Miloradovic V, Topic D, Paunovic D. First clinical comparison of Nobori -Biolimus A9 eluting stents with Cypher- Sirolimus eluting stents: Nobori Core nine months angiographic and one year clinical outcomes. EuroIntervention. 2008 Mar;3(5):574-9. doi: 10.4244/eijv3i5a103. PMID 19608483
- [Background] Iakovou I, Schmidt T, Bonizzoni E, Ge L, Sangiorgi GM, Stankovic G, Airoldi F, Chieffo A, Montorfano M, Carlino M, Michev I, Corvaja N, Briguori C, Gerckens U, Grube E, Colombo A. Incidence, predictors, and outcome of thrombosis after successful implantation of drug-eluting stents. JAMA. 2005 May 4;293(17):2126-30. doi: 10.1001/jama.293.17.2126. PMID 15870416
- [Background] Chevalier B, Silber S, Park SJ, Garcia E, Schuler G, Suryapranata H, Koolen J, Hauptmann KE, Wijns W, Morice MC, Carrie D, van Es GA, Nagai H, Detiege D, Paunovic D, Serruys PW; NOBORI 1 Clinical Investigators. Randomized comparison of the Nobori Biolimus A9-eluting coronary stent with the Taxus Liberte paclitaxel-eluting coronary stent in patients with stenosis in native coronary arteries: the NOBORI 1 trial--Phase 2. Circ Cardiovasc Interv. 2009 Jun;2(3):188-95. doi: 10.1161/CIRCINTERVENTIONS.108.823443. Epub 2009 May 8. PMID 20031715
- [Background] Jain AK, Meredith IT, Lotan C, Rothman MT, Pateraki S; E-Five Investigators. Real-world safety and efficacy of the endeavor zotarolimus-eluting stent: early data from the E-Five Registry. Am J Cardiol. 2007 Oct 22;100(8B):77M-83M. doi: 10.1016/j.amjcard.2007.08.026. PMID 17950836
- [Background] Urban P, Gershlick AH, Guagliumi G, Guyon P, Lotan C, Schofer J, Seth A, Sousa JE, Wijns W, Berge C, Deme M, Stoll HP; e-Cypher Investigators. Safety of coronary sirolimus-eluting stents in daily clinical practice: one-year follow-up of the e-Cypher registry. Circulation. 2006 Mar 21;113(11):1434-41. doi: 10.1161/CIRCULATIONAHA.104.532242. Epub 2006 Mar 13. PMID 16534015
- [Background] Stone GW. SPIRIT IV A Prospective, Randomized Trial Comparing an Everolimus Eluting Stent and a Paclitaxel Eluting Stent in Patients With Coronary Artery Disease One Year Clinical Results. 2009.
- [Background] Grube E, Spirit V registry: one-year follow-up. EuroIntervention 2009; 5
- [Background] Turco MA, Ormiston JA, Popma JJ, Mandinov L, O'Shaughnessy CD, Mann T, McGarry TF, Wu CJ, Chan C, Webster MW, Hall JJ, Mishkel GJ, Cannon LA, Baim DS, Koglin J. Polymer-based, paclitaxel-eluting TAXUS Liberte stent in de novo lesions: the pivotal TAXUS ATLAS trial. J Am Coll Cardiol. 2007 Apr 24;49(16):1676-83. doi: 10.1016/j.jacc.2007.01.069. Epub 2007 Apr 6. PMID 17448368
- [Background] Rodriguez-Granillo GA, Valgimigli M, Garcia-Garcia HM, Ong AT, Aoki J, van Mieghem CA, Tsuchida K, Sianos G, McFadden E, van der Giessen WJ, van Domburg R, de Feyter P, Serruys PW. One-year clinical outcome after coronary stenting of very small vessels using 2.25 mm sirolimus- and paclitaxel-eluting stents: a comparison between the RESEARCH and T-SEARCH registries. J Invasive Cardiol. 2005 Aug;17(8):409-12. PMID 16079445
- [Background] Ong AT, van Domburg RT, Aoki J, Sonnenschein K, Lemos PA, Serruys PW. Sirolimus-eluting stents remain superior to bare-metal stents at two years: medium-term results from the Rapamycin-Eluting Stent Evaluated at Rotterdam Cardiology Hospital (RESEARCH) registry. J Am Coll Cardiol. 2006 Apr 4;47(7):1356-60. doi: 10.1016/j.jacc.2005.05.102. Epub 2006 Mar 20. PMID 16580521
- [Background] Galloe AM, Thuesen L, Kelbaek H, Thayssen P, Rasmussen K, Hansen PR, Bligaard N, Saunamaki K, Junker A, Aaroe J, Abildgaard U, Ravkilde J, Engstrom T, Jensen JS, Andersen HR, Botker HE, Galatius S, Kristensen SD, Madsen JK, Krusell LR, Abildstrom SZ, Stephansen GB, Lassen JF; SORT OUT II Investigators. Comparison of paclitaxel- and sirolimus-eluting stents in everyday clinical practice: the SORT OUT II randomized trial. JAMA. 2008 Jan 30;299(4):409-16. doi: 10.1001/jama.299.4.409. PMID 18230778
- [Background] Kedhi E, Joesoef KS, McFadden E, Wassing J, van Mieghem C, Goedhart D, Smits PC. Second-generation everolimus-eluting and paclitaxel-eluting stents in real-life practice (COMPARE): a randomised trial. Lancet. 2010 Jan 16;375(9710):201-9. doi: 10.1016/S0140-6736(09)62127-9. Epub 2010 Jan 7. PMID 20060578
- [Background] Novack V, Cutlip D, Kleiman N, Pencina M, Mauri L, Yen CH, Berger P, Goldberg S, Kellett M, Waksman R, Hong M, Raizner AE, Cohen DJ. In-hospital and 1-year outcomes among unselected percutaneous coronary intervention patients treated with either sirolimus- or paclitaxel-eluting stents: results from the EVENT (Evaluation of Drug Eluting Stents and Ischemic Events) registry. JACC Cardiovasc Interv. 2009 Aug;2(8):767-75. doi: 10.1016/j.jcin.2009.05.016. PMID 19695546
- [Background] Windecker S, Serruys PW, Wandel S, Buszman P, Trznadel S, Linke A, Lenk K, Ischinger T, Klauss V, Eberli F, Corti R, Wijns W, Morice MC, di Mario C, Davies S, van Geuns RJ, Eerdmans P, van Es GA, Meier B, Juni P. Biolimus-eluting stent with biodegradable polymer versus sirolimus-eluting stent with durable polymer for coronary revascularisation (LEADERS): a randomised non-inferiority trial. Lancet. 2008 Sep 27;372(9644):1163-73. doi: 10.1016/S0140-6736(08)61244-1. Epub 2008 Aug 31. PMID 18765162
- [Background] Silber S, Albertsson P, Aviles FF, Camici PG, Colombo A, Hamm C, Jorgensen E, Marco J, Nordrehaug JE, Ruzyllo W, Urban P, Stone GW, Wijns W; Task Force for Percutaneous Coronary Interventions of the European Society of Cardiology. Guidelines for percutaneous coronary interventions. The Task Force for Percutaneous Coronary Interventions of the European Society of Cardiology. Eur Heart J. 2005 Apr;26(8):804-47. doi: 10.1093/eurheartj/ehi138. Epub 2005 Mar 15. PMID 15769784
- [Background] Shaw LJ, Berman DS, Maron DJ, Mancini GB, Hayes SW, Hartigan PM, Weintraub WS, O'Rourke RA, Dada M, Spertus JA, Chaitman BR, Friedman J, Slomka P, Heller GV, Germano G, Gosselin G, Berger P, Kostuk WJ, Schwartz RG, Knudtson M, Veledar E, Bates ER, McCallister B, Teo KK, Boden WE; COURAGE Investigators. Optimal medical therapy with or without percutaneous coronary intervention to reduce ischemic burden: results from the Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation (COURAGE) trial nuclear substudy. Circulation. 2008 Mar 11;117(10):1283-91. doi: 10.1161/CIRCULATIONAHA.107.743963. Epub 2008 Feb 11. PMID 18268144
- [Background] Safian R.D. and Freed M., Complications. In: The Manual of Interventional Cardiology Jones & Bartlett Publishers, 2001. 381-467
- [Background] Tillmanns H, Waas W, Voss R, Grempels E, Holschermann H, Haberbosch W, Waldecker B. Gender differences in the outcome of cardiac interventions. Herz. 2005 Aug;30(5):375-89. doi: 10.1007/s00059-005-2716-3. English, German. PMID 16132240
- [Background] Berger JS, Elliott L, Gallup D, Roe M, Granger CB, Armstrong PW, Simes RJ, White HD, Van de Werf F, Topol EJ, Hochman JS, Newby LK, Harrington RA, Califf RM, Becker RC, Douglas PS. Sex differences in mortality following acute coronary syndromes. JAMA. 2009 Aug 26;302(8):874-82. doi: 10.1001/jama.2009.1227. PMID 19706861
- [Background] Briguori C, Airoldi F, Chieffo A, Carlino M, Montorfano M, Colombo A. Renal function and drug-eluting stent. Int J Cardiol. 2010 Jun 25;142(1):92-4. doi: 10.1016/j.ijcard.2008.11.138. Epub 2009 Jan 15. PMID 19147241
- [Background] Latif F, Kleiman NS, Cohen DJ, Pencina MJ, Yen CH, Cutlip DE, Moliterno DJ, Nassif D, Lopez JJ, Saucedo JF; EVENT Investigators. In-hospital and 1-year outcomes among percutaneous coronary intervention patients with chronic kidney disease in the era of drug-eluting stents: a report from the EVENT (Evaluation of Drug Eluting Stents and Ischemic Events) registry. JACC Cardiovasc Interv. 2009 Jan;2(1):37-45. doi: 10.1016/j.jcin.2008.06.012. PMID 19463396
- [Background] Rosenblum MA, Robbins MJ, Farkouh ME, Winston JA, Kim MC. Diminished benefits of drug-eluting stents versus bare metal stents in patients with severe renal insufficiency. Nephron Clin Pract. 2009;113(3):c198-202. doi: 10.1159/000232602. Epub 2009 Aug 12. PMID 19672119
- [Background] Mehilli J, Dibra A, Kastrati A, Pache J, Dirschinger J, Schomig A; Intracoronary Drug-Eluting Stenting to Abrogate Restenosis in Small Arteries (ISAR-SMART 3) Study Investigators. Randomized trial of paclitaxel- and sirolimus-eluting stents in small coronary vessels. Eur Heart J. 2006 Feb;27(3):260-6. doi: 10.1093/eurheartj/ehi721. Epub 2006 Jan 9. PMID 16401670
- [Background] Park SW, Lee CW, Hong MK, Kim JJ, Cho GY, Nah DY, Park SJ. Randomized comparison of coronary stenting with optimal balloon angioplasty for treatment of lesions in small coronary arteries. Eur Heart J. 2000 Nov;21(21):1785-9. doi: 10.1053/euhj.1999.1947. PMID 11052843
- [Background] Ortolani P, Marzocchi A, Marrozzini C, Palmerini T, Saia F, Taglieri N, Aquilina M, Baldazzi F, Silenzi S, Cooke RM, Reggiani ML, Branzi A. Randomized comparative trial of a thin-strut bare metal cobalt-chromium stent versus a sirolimus-eluting stent for coronary revascularization. Catheter Cardiovasc Interv. 2007 May 1;69(6):790-8. doi: 10.1002/ccd.21011. PMID 17290437
- [Background] Tanimoto S, Daemen J, Serruys PW. Update on stents: recent studies on the TAXUS stent system in small vessels. Vasc Health Risk Manag. 2007;3(4):481-90. PMID 17969378
- [Background] Elezi S, Kastrati A, Pache J, Wehinger A, Hadamitzky M, Dirschinger J, Neumann FJ, Schomig A. Diabetes mellitus and the clinical and angiographic outcome after coronary stent placement. J Am Coll Cardiol. 1998 Dec;32(7):1866-73. doi: 10.1016/s0735-1097(98)00467-7. PMID 9857865
- [Background] Stettler C, Allemann S, Egger M, Windecker S, Meier B, Diem P. Efficacy of drug eluting stents in patients with and without diabetes mellitus: indirect comparison of controlled trials. Heart. 2006 May;92(5):650-7. doi: 10.1136/hrt.2005.070698. Epub 2005 Oct 26. PMID 16251229
- [Background] Boccara F, Teiger E, Cohen A. Role of drug eluting stents in diabetic patients. Heart. 2006 May;92(5):579-81. doi: 10.1136/hrt.2005.082172. Epub 2006 Jan 31. PMID 16449508
- [Background] Sukhija R, Mehta JL, Sachdeva R. Present status of coronary bifurcation stenting. Clin Cardiol. 2008 Feb;31(2):63-6. doi: 10.1002/clc.20177. PMID 17763364
- [Background] Kim YH, Park SW, Lee SW, Park DW, Yun SC, Lee CW, Hong MK, Kim HS, Ko JK, Park JH, Lee JH, Choi SW, Seong IW, Cho YH, Lee NH, Kim JH, Chun KJ, Park SJ; Long-DES-II Study Investigators. Sirolimus-eluting stent versus paclitaxel-eluting stent for patients with long coronary artery disease. Circulation. 2006 Nov 14;114(20):2148-53. doi: 10.1161/CIRCULATIONAHA.106.666396. Epub 2006 Oct 23. PMID 17060388
- [Background] Hannan EL, Wu C, Walford G, Culliford AT, Gold JP, Smith CR, Higgins RS, Carlson RE, Jones RH. Drug-eluting stents vs. coronary-artery bypass grafting in multivessel coronary disease. N Engl J Med. 2008 Jan 24;358(4):331-41. doi: 10.1056/NEJMoa071804. PMID 18216353
- [Background] Nakamura S, Nakamura S, Ogawa H, Bae JH, HansCahyadi Y, Udayachalerm W, DTresukosol D, Tansuphaswadikul S, Drug-eluting stents for the treatment of left main coronary artery disease with sirolimus, paclitaxel, zotarolimus, BiolimusA9, EPC capture and everolimus-eluting stent: multicenter registry in Asia (Oral Contributions Georgia World Congress Center, Room B315 Monday, March 15, 2010, 2:00 p.m.-2:12 p.m.). J Am Coll Cardiol 2010;55
- [Background] Lotan C, Almagor Y, Kuiper K, Suttorp MJ, Wijns W. Sirolimus-eluting stent in chronic total occlusion: the SICTO study. J Interv Cardiol. 2006 Aug;19(4):307-12. doi: 10.1111/j.1540-8183.2006.00151.x. PMID 16881976
- [Background] Rahel BM, Suttorp MJ, Laarman GJ, Kiemeneij F, Bal ET, Rensing BJ, Ernst SM, ten Berg JM, Kelder JC, Plokker HW. Primary stenting of occluded native coronary arteries: final results of the Primary Stenting of Occluded Native Coronary Arteries (PRISON) study. Am Heart J. 2004 May;147(5):e22. doi: 10.1016/j.ahj.2003.11.023. PMID 15131557
- [Background] Suttorp MJ, Laarman GJ, Rahel BM, Kelder JC, Bosschaert MA, Kiemeneij F, Ten Berg JM, Bal ET, Rensing BJ, Eefting FD, Mast EG. Primary Stenting of Totally Occluded Native Coronary Arteries II (PRISON II): a randomized comparison of bare metal stent implantation with sirolimus-eluting stent implantation for the treatment of total coronary occlusions. Circulation. 2006 Aug 29;114(9):921-8. doi: 10.1161/CIRCULATIONAHA.106.613588. Epub 2006 Aug 14. PMID 16908768
- [Background] Nakamura S, Nakamura S, Ogawa H, Bae JH, HansCahyadi Y, Udayachalerm W, DTresukosol D, Tansuphaswadikul S, Drug-eluting stents for the treatment of chronic total occlusion: a comparison with sirolimus, paclitaxel, zotarolimus, BiolimusA9, EPC capture and everolimus-eluting stent: multicenter registry in Asia (Poster Contributions Georgia World Congress Center, Hall B5 Monday, March 15, 2010, 9:30 a.m.-10:30 a.m. ). J Am Coll Cardiol 2010;55.
- [Background] Hamm CW, Braunwald E. A classification of unstable angina revisited. Circulation. 2000 Jul 4;102(1):118-22. doi: 10.1161/01.cir.102.1.118. PMID 10880424
- [Background] Braunwald E. Unstable angina. A classification. Circulation. 1989 Aug;80(2):410-4. doi: 10.1161/01.cir.80.2.410. No abstract available. PMID 2752565
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] TIMI Study Group. The Thrombolysis in Myocardial Infarction (TIMI) trial. Phase I findings. N Engl J Med. 1985 Apr 4;312(14):932-6. doi: 10.1056/NEJM198504043121437. No abstract available. PMID 4038784